CLINICAL TRIAL: NCT00984724
Title: Reducing Tobacco Related Health Disparities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009-0372; 1R01CA141613-01 (NIH); NCI-2011-00289 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-09-23; First posted 2009-09-25 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Smoking Cessation; Smoking
Keywords: Smoking; Motivation and Problem Solving; MAPS; Low Income Smokers; HCHD community clinics; Telephone-based counseling
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Standard Treatment (Experimental): Standard Treatment (ST): Mailed Packet with standard self-help materials; ST delivered a total of 4 times (at Baseline, 6, 12, and 18 months). Referral to Quitline.
  Interventions: Behavioral: Standard Treatment (ST); Behavioral: Quitline
- MAPS-6 (Experimental): Standard Treatment (ST) plus 6 proactive telephone counseling sessions; ST delivered 4 times (at Baseline, 6, 12, and 18 months). 6 MAPS proactive telephone counseling sessions over 2-year period.
  Interventions: Behavioral: Standard Treatment (ST); Behavioral: Telephone Counseling; Behavioral: Quitline
- MAPS-12 (Experimental): Standard Treatment (ST) plus 12 proactive telephone counseling sessions; ST delivered 4 times (at Baseline, 6, 12, and 18 months). 12 MAPS proactive telephone counseling sessions over 2-year period. Referral to Quitline.
  Interventions: Behavioral: Standard Treatment (ST); Behavioral: Telephone Counseling; Behavioral: Quitline
- Standard Treatment + NRT (Experimental): Standard Treatment (ST): Mailed Packet with standard self-help materials; ST delivered a total of 4 times (at Baseline, 6, 12, and 18 months). Nicotine replacement therapy (NRT) consisting of 300 pieces of nicotine gum issued at baseline visit.
  Interventions: Behavioral: Standard Treatment (ST); Behavioral: Quitline; Behavioral: Nicotine Replacement Therapy (NRT)
- MAPS-6 + NRT (Experimental): Standard Treatment (ST) plus 6 proactive telephone counseling sessions; delivered 4 times (at Baseline, 6, 12, and 18 months). 6 MAPS proactive telephone counseling sessions over 2-year period. Referral to Quitline. Nicotine replacement therapy (NRT) consisting of 300 pieces of nicotine gum issued at baseline visit.
  Interventions: Behavioral: Standard Treatment (ST); Behavioral: Telephone Counseling; Behavioral: Quitline; Behavioral: Nicotine Replacement Therapy (NRT)
- MAPS-12 + NRT (Experimental): Standard Treatment (ST) plus 12 proactive telephone counseling sessions; ST delivered 4 times (at Baseline, 6, 12, and 18 months). 12 MAPS proactive telephone counseling sessions over 2-year period. Referral to Quitline. Nicotine replacement therapy (NRT) consisting of 300 pieces of nicotine gum issued at baseline visit.
  Interventions: Behavioral: Standard Treatment (ST); Behavioral: Telephone Counseling; Behavioral: Quitline; Behavioral: Nicotine Replacement Therapy (NRT)

INTERVENTIONS:
Behavioral: Standard Treatment (ST) — Mailing of packet of materials including a letter referring smokers to the Texas Quitline, nicotine replacement therapy when participants are ready to quit and standard self-help materials; ST delivered a total of 4 times (at Baseline, 6, 12, and 18 months).
Behavioral: Telephone Counseling — MAPS-6: 6 MAPS proactive telephone counseling sessions delivered over a 2-year period
  MAPS-12: 12 MAPS proactive telephone counseling sessions over a 2-year period
  Arms: MAPS-12; MAPS-12 + NRT; MAPS-6; MAPS-6 + NRT
Behavioral: Quitline — Letter referring participants to a Quitline providing quit smoking services.
Behavioral: Nicotine Replacement Therapy (NRT) — 300 pieces of nicotine gum issued at baseline visit.
  Arms: MAPS-12 + NRT; MAPS-6 + NRT; Standard Treatment + NRT

SUMMARY:
The goal of this research study is to learn the effectiveness of telephone-based counseling on helping smokers change their smoking patterns.

DETAILED DESCRIPTION:
Researchers want to learn if telephone counseling can help smokers change their smoking patterns, when combined with other interventions.

Study Groups:

During the first (baseline) visit, you will be randomly assigned (as in a throw of the dice) to 1 of 4 study groups. The first group will receive free self-help materials, and a referral to the Quitline. The Quitline provides free quit smoking services to eligible callers. The second group will receive free self-help materials, a referral to the Quitline, and 300 pieces of nicotine gum at baseline. The third group will receive free self-help materials, a referral to the Quitline, and 4 telephone counseling sessions over the next month. The fourth group will receive free self-help materials, a referral to the Quitline, 4 telephone counseling sessions over the next month, and 300 pieces of nicotine gum at baseline.

Study Visits:

If you choose to take part in this study, you will visit MD Anderson twice. Your first visit is the "baseline" visit when you enter the study and your final visit is the "follow-up" visit, which is 1 month after baseline.

Study Tests:

The following tests and procedures will be performed at the study visits:

* You will be asked to complete some questionnaires that will include questions about your feelings, moods, and smoking status. These will take 60 to 90 minutes to complete.
* You will have your height, weight, and waistline measured.
* You will complete a breath test to help estimate (guess) the amount of cigarette smoke you inhale. The breath test uses a disposable cardboard tube that is attached to the machine, and you blow a long, slow, steady breath into it.
* You will have saliva samples collected for cotinine tests. To collect the saliva, you will be asked to put a small piece of cotton in your mouth for a few minutes. These samples will be used to measure the amount of cotinine in your saliva. Cotinine is a chemical released in your body when it breaks down nicotine.

All participants will be contacted by mail or telephone throughout the length of the study. You may be contacted by mail, telephone, and/or e-mail during the study and follow-up, to be given reminders of clinic visits. You will be asked to provide the names and contact information for family and/or friends for the study staff to contact if the study staff has trouble reaching you.

Genetic Testing:

As part of this study, you will be asked to provide a saliva sample that will be collected at the first visit. To collect the saliva sample, you will be spitting into a container. Researchers will perform genetic tests with these samples to look for genes that control the production and use of neurotransmitters, naturally occurring chemical messengers in the brain. People with certain genes may have a more difficult time quitting smoking, because of the way nicotine affects these chemicals. The saliva sample will be stored in a biorepository at MD Anderson for use in future research related to nicotine addiction, smoking, and/or cancer.

Your saliva sample will be placed in a bank of biological samples and data that is available to researchers conducting research related to cancer or nicotine dependence.

Before your saliva sample can be used for research, the people doing the research must get specific approval from the Institutional Review Board (IRB) of M. D. Anderson. The IRB is a committee made up of doctors, researchers, and members of the community. The IRB is responsible for protecting the participants involved in research studies and making sure all research is done in a safe and ethical manner. All research done at MD Anderson, including research involving your saliva sample from this bank, must first be approved by the IRB.

Your samples will be given a code number. No identifying information will be directly linked to your samples. Only the researcher in charge of the bank will have access to the code numbers and be able to link the samples to you. Other researchers using your samples will not be able to link this data to you.

Genetic information obtained will not be provided to you.

Telephone Counseling:

The telephone counseling sessions will be digitally recorded. The recordings, if not destroyed, may be kept for use in future research studies. The recordings will be used to help the researchers make sure that the counselors are following the correct procedures and may be used in the future to help the investigators better understand or improve the counseling treatment. No one but the study investigators and their staff will be allowed to view or listen to the recordings, and the identity of the participants will be kept strictly confidential. Your study identification number will be stated by the counselor at the beginning of the taped session. The recordings are stored digitally, encrypted, and password protected.

This is an investigational study. The nicotine gum used in this study is approved by the FDA. Up to 100 smokers will take part in this research study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. HCHD Patient or is at or below 200% of the poverty guideline
2. 18 years of age or older
3. Current smoker
4. History of at least one cigarette per day for the past year
5. Not ready to quit in the next 30 days
6. Valid home address
7. Functioning telephone number
8. Can speak, read, and understand English
9. Register "5" or more on a carbon monoxide breath test

Exclusion Criteria:

1. Other household members enrolled in this study
2. Enrolled in any other smoking study during the past 90 days
3. Scores below the 6th grade literacy level on the Rapid Estimate of Adult Literacy in Medicine (REALM)
4. Regular use of tobacco products other than cigarettes
5. Pregnancy or lactation
6. Active substance dependence (exclusive of nicotine dependence)
7. Use of bupropion or nicotine products

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 639 (Actual)
Dates: Start 2011-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Tobacco Abstinence | 24 months
  Prolonged abstinence refers to abstinence beginning with initiation of the intervention and including a grace period. Prolonged abstinence measure utilizes the Society for Research on Nicotine and Tobacco's recommendation for determining relapse (i.e., 7 consecutive days of smoking or smoking in each of 2 consecutive weeks). Abstinence at all follow-ups will be biochemically verified using a carbon monoxide level of <10ppm. Saliva samples collected for cotinine tests at the baseline and 24 month follow-up visits. Saliva samples analyzed for cotinine, a metabolic byproduct of nicotine that provides an estimate of nicotine consumption. A saliva cotinine level of <20 ng/ml considered as abstinent.

CONTACTS AND LOCATIONS:
Overall Officials: Larkin L. Strong, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Theodoulou A, Chepkin SC, Ye W, Fanshawe TR, Bullen C, Hartmann-Boyce J, Livingstone-Banks J, Hajizadeh A, Lindson N. Different doses, durations and modes of delivery of nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2023 Jun 19;6(6):CD013308. doi: 10.1002/14651858.CD013308.pub2. PMID 37335995
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org